CLINICAL TRIAL: NCT05019521
Title: A Phase 2, Double-Masked, Placebo-Controlled, Dose Range Finding Study of Danicopan (ALXN2040) in Patients With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: A Study of Danicopan in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALXN2040-GA-201; 2021-001198-22 (EudraCT Number)
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Geographic Atrophy
Keywords: Geographic Atrophy; GA; Danicopan; ALXN2040; Complement Inhibition; AMD
MeSH Terms: conditions — Geographic Atrophy | interventions — danicopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking of treatment allocation will be observed until Week 104.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Danicopan: 100 mg (Experimental): Participants will receive danicopan 100 mg bid during the masked Treatment Period. Once the optimal dose is identified, participants who have at least 52 weeks of treatment will be switched to the optimal dose for the remainder of the study.
  Interventions: Drug: Danicopan
- Danicopan: 200 mg (Experimental): Participants will receive danicopan 200 mg bid during the masked Treatment Period. Once the optimal dose is identified, participants who have at least 52 weeks of treatment will be switched to the optimal dose for the remainder of the study.
  Interventions: Drug: Danicopan
- Danicopan: 400 mg (Experimental): Participants will receive danicopan 400 mg qd during the masked Treatment Period. Once the optimal dose is identified, participants who have at least 52 weeks of treatment will be switched to the optimal dose for the remainder of the study.
  Interventions: Drug: Danicopan
- Placebo (Placebo Comparator): Participants will receive matching placebo and will be re-randomized to one of the active treatment groups at Week 52, or to the optimal dose, if already identified.
  Interventions: Drug: Danicopan; Drug: Placebo

INTERVENTIONS:
Drug: Danicopan — Oral tablet.
  Other Names: ALXN2040
Drug: Placebo — Oral tablet.
  Arms: Placebo

SUMMARY:
This is a dose finding study designed to evaluate the efficacy, safety, and pharmacokinetics of danicopan in participants with GA secondary to AMD. The study consists of a Screening Period of up to 6 weeks, a 104-week masked Treatment Period, followed by a 30-day Follow-up after the last dose. This study will have 4 treatments arms: 100 milligrams (mg) twice daily (bid), 200 mg bid, 400 mg once daily (qd), and matching placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Vaccination for Neisseria meningitidis.
* Capable of giving signed informed consent.
* Presentation of GA secondary to AMD in at least 1 eye
* The entire GA lesion must be > 1 μm outside of the foveal center

Key Exclusion Criteria:

* GA in the study eye due to cause other than AMD.
* Have previously received intravitreal anti-vascular endothelial growth factor injections in study eye for intraocular vascular disease.
* Have previously received any stem cell/gene therapy for any ophthalmological condition in either eye.
* Use of any investigational medicinal product (ie, participation in interventional clinical studies for any ophthalmic indications) or use of any regulatory approved treatment for GA in the study eye regardless of route of administration within the last 3 months or 5 half-lives of the last dose of the investigational or commercial product (whichever is longer).
* Presence of active ocular diseases in the study eye that in the opinion of the Investigator compromises or confounds visual function or interferes with study assessments.
* Known or suspected complement deficiency.
* History or presence of any medical or psychological condition that, in the opinion of the Principal Investigator, would make the patient inappropriate for the study.
* Hypersensitivity to fluorescein sodium for injection, the investigational drug (danicopan) or any of its excipients.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2025-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (114):
- United States (48):
  - Research Site, Phoenix, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Encino, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Pasadena, California
  - Research Site, Sacramento, California
  - Research Site, San Mateo, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Longmont, Colorado
  - Research Site, Waterford, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Naples, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Augusta, Georgia
  - Research Site, New Albany, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Hagerstown, Maryland
  - Research Site, Rosedale, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Springfield, Massachusetts
  - Research Site, Southaven, Mississippi
  - Research Site, Reno, Nevada
  - Research Site, Teaneck, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Springfield, Oregon
  - Research Site, Kingston, Pennsylvania
  - Research Site, Monroeville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Ladson, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Austin, Texas
  - Research Site, Bellaire, Texas
  - Research Site, Conroe, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Southlake, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Lynchburg, Virginia
- Australia (7):
  - Research Site, Adelaide
  - Research Site, Albury
  - Research Site, East Melbourne
  - Research Site, Hurstville
  - Research Site, Parramatta
  - Research Site, Strathfield
  - Research Site, Sydney
- Czechia (2):
  - Research Site, Pardubice
  - Research Site, Prague
- France (9):
  - Research Site, Créteil
  - Research Site, Écully
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Strasbourg
- Germany (16):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Mainz A. Rhein
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Münster
  - Research Site, Neubrandenburg
  - Research Site, Regensburg
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Würzburg
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Pécs
- Italy (5):
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Naples
  - Research Site, Roma
- Japan (3):
  - Research Site, Fukushima
  - Research Site, Kita-gun
  - Research Site, Osaka
- Research Site, Riga, Latvia
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Žilina
- South Korea (5):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seoul
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Córdoba
  - Research Site, Majadahonda
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Zaragoza
- United Kingdom (5):
  - Research Site, Bristol
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Southampton

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN2040-GA-201&attachmentIdentifier=58bd7a43-4152-40f6-8310-92f7a766fd0d&fileName=ALXN2040-GA-201_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included 104-week Masked Treatment Period (Masked Placebo-controlled [Primary Evaluation Period; up to 52 weeks] and Masked Active Treatment [Secondary Evaluation Period; Week 52 to Week 104]). As prespecified, data were collected and reported for the participants. Therefore, the 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated.
Pre-assignment Details: For standardization purposes, the primary and secondary efficacy analyses were measured in the pre-specified study eye per individual participant. In this study, ocular assessments were performed in both eyes at Screening. The eye that met all eligibility criteria was designated as the study eye and the other eye was used as the fellow eye. If both eyes were eligible, the right eye was designated as the study eye.
Groups:
- Danicopan 100 mg BID: Participants received danicopan 100 milligrams (mg) twice daily (BID) during the 104-week Masked Treatment Period.
- Danicopan 200 mg BID: Participants received danicopan 200 mg BID during the 104-week Masked Treatment Period.
- Danicopan 400 mg QD: Participants received danicopan 400 mg once daily (QD) during the 104-week Masked Treatment Period.
- Placebo: Participants received matching placebo and were re-randomized to one of the active treatment groups at Week 52.
- Placebo - Danicopan 100 mg BID: Participants who received placebo during the primary evaluation period (up to Week 52), were re-randomized to receive danicopan 100 mg BID for the remainder of the study.
- Placebo - Danicopan 200 mg BID: Participants who received placebo during the primary evaluation period (up to Week 52), were re-randomized to receive danicopan 200 mg BID for the remainder of the study.
- Placebo - Danicopan 400 mg QD: Participants who received placebo during the primary evaluation period (up to Week 52), were re-randomized to receive danicopan 400 mg QD for the remainder of the study.
Period: Primary Evaluation Period (52 Weeks)
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Started | 93 | 91 | 91 | 90 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 93 | 91 | 91 | 90 | 0 | 0 | 0
Completed | 73 | 67 | 73 | 70 | 0 | 0 | 0
Not Completed | 20 | 24 | 18 | 20 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 9 | 8 | 4 | 0 | 0 | 0
Not completed — Investigator's Discretion | 1 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 13 | 6 | 9 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 3 | 0 | 0 | 0
Not completed — Liver abnormalities meeting Hy's Law criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Than Specified | 3 | 0 | 3 | 2 | 0 | 0 | 0
Period: Secondary Evaluation Period (52 Weeks)
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Started | 73 | 67 | 73 | 0 | 24 | 23 | 23
Received at Least 1 Dose of Study Drug | 73 | 67 | 73 | 0 | 24 | 23 | 23
Completed | 15 | 14 | 11 | 0 | 5 | 2 | 3
Not Completed | 58 | 53 | 62 | 0 | 19 | 21 | 20
Not completed — Adverse Event | 2 | 3 | 2 | 0 | 0 | 0 | 3
Not completed — Investigator's Discretion | 1 | 2 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 5 | 2 | 2
Not completed — Lack of Efficacy | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Liver abnormalities meeting Hy's Law criteria | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other Than Specified | 3 | 1 | 3 | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 49 | 45 | 53 | 0 | 13 | 17 | 14

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose (full or partial) of study drug grouped by randomized treatment group. As prespecified, data were collected and reported for the participants. Therefore, the 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated.
Groups:
- Danicopan 100 mg BID: Participants received danicopan 100 mg BID during the 104-week Masked Treatment Period.
- Danicopan 400 mg QD: Participants received danicopan 400 mg QD during the 104-week Masked Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Total
Number analyzed (Participants) | 93 | 91 | 91 | 90 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.0 (7.20) | 76.0 (7.24) | 77.8 (7.52) | 77.8 (6.75) | 77.1 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 58 | 64 | 61 | 251
  Male | 25 | 33 | 27 | 29 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 4 | 6 | 15
  Not Hispanic or Latino | 75 | 81 | 77 | 75 | 308
  Unknown or Not Reported | 14 | 9 | 10 | 9 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 1 | 3 | 3 | 9
  Race: Black or African American | 0 | 0 | 0 | 1 | 1
  Race: White | 77 | 81 | 78 | 76 | 312
  Race: Not Reported | 11 | 6 | 6 | 6 | 29
  Race: Unknown | 3 | 3 | 4 | 2 | 12
  Race: Other | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change From Baseline to Week 52 in the Square Root (Sqrt) of Total Geographic Atrophy (GA) Lesion Area in the Study Eye as Measured by Fundus Autofluorescence (FAF)
Description: FAF provides high-contrast retinal images particularly valuable for the detection of atrophic areas. FAF images of the study eye were taken and sent to the reading center for total GA lesion area measurement. The total GA lesion area (square millimeter [mm^2]) was transformed into sqrt (millimeter [mm]). Greater area affected means a worse outcome than smaller area affected. The rate of change from Baseline (mm/year) for each treatment group was estimated based on the coefficients for time and the interaction of time and treatment from the mixed models for repeated measures (MMRM). MMRM analysis included the change from Baseline at post-baseline visit in the sqrt GA lesion area as dependent variable.
Time Frame: Baseline, Week 52
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) who had any post-baseline FAF GA lesion area data at the Week 52 analysis. As prespecified, data were collected and reported for the participants. Therefore, the 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated.
Measure: Least Squares Mean (Standard Error); unit: mm/year
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo
Number analyzed (Participants) | 65 | 62 | 70 | 66
mm/year | 0.465 (0.0289) | 0.391 (0.0306) | 0.443 (0.0301) | 0.406 (0.0304)
Statistical Analysis 1: Comparison: Danicopan 100 mg BID vs Placebo; Test type: Superiority; p = 0.9205, Mixed Models Analysis; Least square (LS) mean difference = 0.058, 90% CI 2-sided [-0.010 to 0.126], Standard Error of Mean 0.0413
Statistical Analysis 2: Comparison: Danicopan 200 mg BID vs Placebo; Test type: Superiority; p = 0.9205, Mixed Models Analysis; LS mean difference = -0.016, 90% CI 2-sided [-0.086 to 0.055], Standard Error of Mean 0.0425
Statistical Analysis 3: Comparison: Danicopan 400 mg QD vs Placebo; Test type: Superiority; p = 0.9205, Mixed Models Analysis; LS mean difference = 0.037, 90% CI 2-sided [-0.033 to 0.106], Standard Error of Mean 0.0422

2. Secondary Outcome: Change From Baseline to Week 104 in the Sqrt of the Total GA Lesion Area in the Study Eye as Measured by FAF
Description: FAF provides high-contrast retinal images particularly valuable for the detection of atrophic areas. FAF images of the study eye were taken and sent to the reading center for total GA lesion area measurement. The total GA lesion area (mm^2) was transformed into sqrt (mm). Greater area affected means a worse outcome than smaller area affected.
Time Frame: Baseline, Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline visit and post-baseline (Week 104) visit FAF GA lesion area data. As prespecified, data were collected and reported for the participants. Therefore, the 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 18 | 13 | 18 | 6 | 4 | 4
mm | 0.892 (0.4545) | 0.705 (0.3831) | 0.859 (0.3468) | 0.668 (0.4866) | 0.585 (0.1396) | 0.787 (0.1858)

3. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in the Total GA Lesion Area in the Study Eye as Measured by FAF
Description: FAF provides high-contrast retinal images particularly valuable for the detection of atrophic areas. FAF images of the study eye were taken and sent to the reading center for total GA lesion area (mm^2) measurement. Greater area affected means a worse outcome than smaller area affected.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit FAF GA lesion area data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 65 | 62 | 70 | 66 | 24 | 20 | 22
mm^2
  Change at Week 52 | 2.347 (1.2972) | 2.044 (1.2280) | 2.274 (1.4482) | 2.057 (1.2016) | 1.887 (1.1212) | 1.716 (0.9095) | 2.553 (1.3938)
  Change at Week 104: number analyzed (Participants) | 18 | 13 | 18 | 0 | 6 | 4 | 4
  Change at Week 104 | 4.311 (2.8803) | 3.223 (2.3784) | 4.504 (2.1300) |  | 3.309 (2.5878) | 3.653 (2.3125) | 5.098 (1.8250)

4. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Macular Ellipsoid Zone (EZ) Total Attenuation in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by Spectral-domain Optical Coherence Tomography (SD-OCT)
Description: Photoreceptor loss was assessed by measuring the percent of macular EZ total attenuation using SD-OCT. The EZ was considered to be formed mainly by mitochondria within the ellipsoid layer of the outer portion of the inner segments of the photoreceptors. In SD-OCT, decreases in the integrity and intensity of the EZ have been correlated with the reduction in cone photoreceptors and retinal sensitivity in retinal degenerative diseases. Lower increase in percentage means a better outcome. Higher increase in percentage means a worse outcome.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit SD-OCT data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: percentage of EZ total attenuation
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of EZ total attenuation
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 64 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 8.70 (4.681) | 7.48 (4.226) | 8.66 (4.633) | 7.50 (4.814) | 6.03 (3.147) | 7.74 (4.469) | 8.77 (6.206)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 16 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 13.54 (7.664) | 11.72 (7.976) | 15.27 (6.156) |  | 10.81 (6.514) | 12.65 (5.163) | 14.76 (6.672)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 6.31 (3.642) | 5.53 (3.665) | 6.96 (4.684) | 7.87 (4.790) | 7.31 (4.898) | 7.26 (4.164) | 8.94 (5.205)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 12.80 (7.605) | 9.48 (5.396) | 14.05 (9.509) |  | 11.82 (9.719) | 12.34 (5.174) | 14.19 (3.223)
  Both Eyes Combined: Change at Week 52 | 13.77 (7.285) | 11.27 (6.892) | 14.94 (8.335) | 14.02 (8.564) | 12.17 (7.625) | 13.43 (7.072) | 16.55 (10.412)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 22.18 (15.324) | 17.17 (13.337) | 28.51 (12.937) |  | 20.65 (15.245) | 22.53 (7.748) | 28.95 (7.702)

5. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Macular EZ Partial Attenuation in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: Photoreceptor degradation was assessed by measuring the percent of macular EZ partial attenuation using SD-OCT. The EZ was considered to be formed mainly by mitochondria within the ellipsoid layer of the outer portion of the inner segments of the photoreceptors. In SD-OCT, decreases in the integrity and intensity of the EZ have been correlated with the reduction in cone photoreceptors and retinal sensitivity in retinal degenerative diseases. Lower increase in percentage means a better outcome. Higher increase in percentage means a worse outcome.
Time Frame: Baseline, Week 52 and Week 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of EZ partial attenuation
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of EZ partial attenuation
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 64 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 6.42 (4.917) | 5.15 (3.806) | 6.63 (4.599) | 5.65 (4.365) | 4.00 (3.423) | 5.54 (4.089) | 7.49 (4.946)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 16 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 12.48 (7.290) | 8.06 (6.728) | 13.87 (7.495) |  | 7.75 (4.677) | 10.55 (7.536) | 10.56 (6.122)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 5.74 (4.531) | 4.28 (3.646) | 5.61 (4.987) | 6.31 (4.370) | 4.90 (3.399) | 5.83 (4.616) | 8.15 (4.563)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 11.09 (6.771) | 7.87 (5.927) | 13.79 (9.773) |  | 6.20 (6.897) | 11.52 (8.433) | 13.48 (3.926)
  Both Eyes Combined: Change at Week 52 | 11.10 (8.110) | 8.10 (5.976) | 11.69 (8.277) | 10.90 (7.617) | 8.11 (5.784) | 10.10 (6.989) | 14.60 (8.644)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 19.85 (14.357) | 12.67 (10.789) | 26.92 (14.542) |  | 12.92 (10.399) | 19.77 (11.361) | 24.04 (8.185)

6. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Outer Nuclear Layer (ONL) - Retinal Pigment Epithelium (RPE) Mean Central 1 mm Subfield Thickness in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The ONL - RPE mean central 1 mm subfield thickness refers to the average thickness of the retinal layers between the ONL and RPE measured within a 1 mm radius from the foveal center (the central point of the retina).
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment) with both baseline and post-baseline (Week 52 and Week 104) visit ONL-RPE mean central 1 mm subfield thickness data. As prespecified, data were collected and reported for participants. Hence, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: micrometers (µm)
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
micrometers (µm)
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | -4.60 (13.366) | -4.48 (13.398) | -4.86 (13.345) | -3.10 (10.666) | -0.51 (10.404) | -2.53 (8.417) | -6.41 (12.496)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | -12.63 (23.455) | -10.01 (29.953) | -12.47 (23.648) |  | -22.77 (38.733) | -14.72 (14.931) | -12.76 (15.206)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | -7.83 (13.457) | -4.65 (12.206) | -7.63 (15.236) | -7.63 (15.088) | -4.69 (13.097) | -9.01 (17.029) | -9.39 (15.478)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | -13.84 (25.155) | -12.00 (6.459) | -16.53 (25.363) |  | -14.28 (14.915) | -26.53 (10.412) | -26.32 (18.045)
  Both Eyes Combined: Change at Week 52 | -11.16 (16.448) | -7.77 (18.785) | -11.75 (21.771) | -9.55 (20.028) | -4.60 (19.446) | -9.57 (19.250) | -14.70 (20.919)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | -22.29 (31.682) | -17.78 (28.793) | -28.34 (39.848) |  | -34.67 (50.039) | -35.94 (25.831) | -39.08 (32.217)

7. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in ONL-RPE Mean Central Macular 2 mm Subfield Thickness in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The ONL - RPE mean central macular 2 mm subfield thickness refers to the thickness of the retina in the central part of the macula, specifically within a 2 mm radius.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment) with both baseline and post-baseline (Week 52 and Week 104) visit ONL-RPE mean central macular 2 mm thickness data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below= number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
µm
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | -7.42 (7.354) | -6.56 (9.960) | -8.04 (8.589) | -7.25 (7.219) | -4.85 (6.749) | -7.53 (6.631) | -9.46 (7.805)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | -17.49 (14.707) | -12.09 (21.562) | -15.47 (11.523) |  | -21.03 (23.221) | -14.62 (6.409) | -19.46 (11.807)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | -8.39 (8.989) | -5.91 (9.783) | -9.01 (8.981) | -7.92 (9.205) | -7.28 (7.784) | -7.04 (7.522) | -9.32 (11.750)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | -14.66 (14.939) | -14.86 (11.321) | -17.60 (10.975) |  | -13.48 (10.615) | -16.20 (4.746) | -20.98 (12.521)
  Both Eyes Combined: Change at Week 52 | -14.33 (11.799) | -10.74 (14.465) | -16.18 (13.333) | -13.83 (12.378) | -11.01 (11.299) | -13.05 (9.983) | -17.56 (14.952)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | -27.07 (19.859) | -21.71 (24.931) | -32.26 (19.723) |  | -32.27 (31.178) | -27.58 (13.280) | -40.44 (23.788)

8. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Ellipsoid Zone (EZ) - (RPE) Macular Volume in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The EZ - RPE macular volume refers to the volume of the retinal tissue between the EZ and the RPE, specifically within the macular region. Changes in EZ-RPE volume indicate the presence or progression of diseases affecting the outer retina.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit EZ-RPE macular volume data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: cubic millimeters (mm^3)
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
cubic millimeters (mm^3)
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 64 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | -0.09 (0.074) | -0.07 (0.047) | -0.09 (0.048) | -0.06 (0.063) | -0.05 (0.063) | -0.06 (0.058) | -0.08 (0.069)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 16 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | -0.18 (0.066) | -0.10 (0.098) | -0.16 (0.089) |  | -0.10 (0.064) | -0.13 (0.107) | -0.12 (0.068)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | -0.08 (0.062) | -0.05 (0.047) | -0.08 (0.059) | -0.07 (0.052) | -0.06 (0.052) | -0.08 (0.052) | -0.08 (0.053)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | -0.16 (0.097) | -0.11 (0.056) | -0.16 (0.122) |  | -0.10 (0.082) | -0.13 (0.075) | -0.16 (0.037)
  Both Eyes Combined: Change at Week 52 | -0.15 (0.115) | -0.10 (0.069) | -0.16 (0.089) | -0.13 (0.098) | -0.11 (0.103) | -0.12 (0.082) | -0.15 (0.106)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | -0.29 (0.170) | -0.17 (0.143) | -0.32 (0.174) |  | -0.18 (0.135) | -0.23 (0.133) | -0.28 (0.069)

9. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in EZ-RPE Mean Central 1 mm Subfield Thickness in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The EZ - RPE mean central 1 mm subfield thickness is a measurement of the thickness of the ellipsoid zone, a layer within the retina, in the central 1 mm region. Changes in EZ-RPE thickness indicate damage or dysfunction within the photoreceptors, which is associated with various eye diseases like AMD.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment) with both baseline and post-baseline (Week 52 and Week 104) visit EZ-RPE mean central 1 mm subfield thickness data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below= number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
µm
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | -4.03 (3.888) | -3.48 (4.243) | -3.83 (4.044) | -3.16 (4.466) | -2.40 (2.863) | -3.85 (6.048) | -3.25 (3.944)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | -8.32 (4.050) | -5.70 (5.327) | -6.47 (5.111) |  | -5.82 (4.866) | -6.76 (6.100) | -2.76 (2.737)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | -2.51 (4.076) | -1.93 (3.043) | -3.01 (3.685) | -3.52 (4.738) | -3.51 (4.338) | -3.42 (4.103) | -3.61 (5.753)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | -5.23 (4.879) | -4.26 (3.160) | -5.05 (4.629) |  | -4.10 (7.591) | -3.15 (3.755) | -4.30 (5.902)
  Both Eyes Combined: Change at Week 52 | -6.03 (6.163) | -4.85 (5.035) | -6.55 (5.942) | -6.09 (6.692) | -5.37 (5.864) | -6.53 (7.175) | -6.40 (7.224)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | -11.41 (8.175) | -8.46 (5.799) | -11.18 (7.506) |  | -9.23 (9.970) | -9.28 (7.248) | -7.06 (7.138)

10. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in EZ-RPE Mean Central Macular 2 mm Thickness in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The EZ - RPE mean central macular 2 mm thickness measurement reflects the distance between the outer border of the EZ and the inner border of the RPE layer, typically within a central 2 mm area. Decreased EZ-RPE thickness is an early indicator of disease, such as in dry AMD, where a thinning or loss of the EZ is a hallmark. Changes in EZ-RPE thickness is used to monitor treatment response in conditions like AMD.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment) with both baseline and post-baseline (Week 52 and Week 104) visit EZ-RPE mean central macular 2 mm thickness data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below= number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
µm
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | -3.45 (2.971) | -2.75 (2.633) | -3.20 (2.622) | -2.58 (2.819) | -2.58 (3.012) | -2.70 (3.011) | -2.45 (2.512)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | -7.44 (3.218) | -5.21 (4.657) | -5.46 (3.400) |  | -5.05 (4.337) | -5.56 (3.808) | -3.00 (1.925)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | -2.51 (3.042) | -1.93 (3.082) | -2.76 (3.147) | -3.22 (3.844) | -3.50 (3.502) | -2.97 (3.983) | -3.16 (4.206)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | -5.58 (5.229) | -3.38 (2.564) | -4.89 (5.228) |  | -3.50 (6.461) | -4.05 (5.544) | -3.80 (4.506)
  Both Eyes Combined: Change at Week 52 | -5.46 (4.343) | -4.11 (3.792) | -5.68 (4.637) | -5.27 (5.408) | -5.54 (5.618) | -5.03 (5.235) | -5.23 (5.584)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | -10.96 (7.034) | -7.40 (5.216) | -10.06 (7.266) |  | -7.97 (8.308) | -8.80 (7.525) | -6.80 (5.094)

11. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Central 1 mm Subfield EZ Total Attenuation in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The percentage of total attenuation of the EZ in the central 1 mm subfield is reported.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit SD-OCT data. As prespecified, data were collected and reported for the participants. Therefore, the 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: percentage of EZ total attenuation
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of EZ total attenuation
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 16.73 (16.914) | 15.93 (21.716) | 18.68 (20.417) | 13.69 (16.939) | 11.07 (13.674) | 12.68 (18.176) | 17.48 (18.703)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 22.31 (17.890) | 20.14 (19.616) | 39.81 (26.391) |  | 19.40 (19.132) | 18.21 (23.796) | 19.61 (16.593)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 9.16 (12.800) | 8.33 (16.198) | 12.68 (16.131) | 13.44 (17.791) | 13.33 (23.449) | 12.33 (10.834) | 14.51 (16.785)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 20.59 (15.693) | 13.59 (16.375) | 24.22 (22.988) |  | 10.43 (12.638) | 13.11 (12.384) | 18.81 (17.001)
  Both Eyes Combined: Change at Week 52 | 23.92 (21.961) | 21.82 (27.888) | 30.13 (26.472) | 24.82 (24.477) | 22.27 (27.116) | 22.33 (20.562) | 29.97 (25.421)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 36.13 (29.699) | 28.93 (27.084) | 61.94 (38.776) |  | 28.09 (27.090) | 28.70 (31.841) | 38.42 (27.959)

12. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Central 1 mm Subfield EZ Partial Attenuation in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The percentage of partial attenuation of the EZ in the central 1 mm subfield is reported.
Time Frame: Baseline, Week 52 and Week 104
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of EZ partial attenuation
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of EZ partial attenuation
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 10.31 (13.668) | 8.24 (12.342) | 9.51 (14.020) | 8.67 (13.691) | 6.65 (7.932) | 11.42 (18.493) | 7.92 (12.672)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 24.56 (14.964) | 16.86 (18.793) | 12.57 (16.778) |  | 17.58 (20.152) | 22.86 (18.298) | 4.08 (5.899)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 6.80 (14.277) | 5.39 (9.926) | 7.26 (12.982) | 9.92 (16.529) | 9.62 (12.575) | 9.45 (13.614) | 10.61 (22.125)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 13.35 (18.080) | 9.25 (10.751) | 12.65 (15.581) |  | 14.87 (29.975) | 5.76 (11.374) | 10.38 (18.139)
  Both Eyes Combined: Change at Week 52 | 15.74 (20.909) | 12.06 (15.349) | 16.06 (20.365) | 16.93 (21.887) | 14.79 (17.280) | 18.81 (23.297) | 17.27 (25.273)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 31.92 (29.615) | 22.85 (20.419) | 24.56 (23.689) |  | 29.97 (39.643) | 27.47 (22.597) | 14.46 (17.962)

13. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Central Macular 2 mm Subfield EZ Total Attenuation in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The percentage of total attenuation of the EZ in the central macular 2 mm subfield is reported.
Time Frame: Baseline, Week 52 and Week 104
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of EZ total attenuation
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of EZ total attenuation
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 16.04 (12.199) | 13.61 (13.797) | 16.10 (12.422) | 12.89 (11.554) | 12.66 (11.515) | 11.15 (8.184) | 14.96 (14.456)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 27.98 (14.597) | 23.25 (15.725) | 32.56 (15.265) |  | 21.46 (20.555) | 17.50 (6.271) | 19.63 (7.982)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 9.80 (11.161) | 8.84 (11.049) | 11.54 (11.821) | 13.21 (12.847) | 15.14 (14.786) | 11.79 (10.311) | 12.48 (13.098)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 21.45 (21.023) | 12.76 (9.657) | 22.72 (20.095) |  | 11.59 (13.028) | 18.41 (13.948) | 16.20 (13.464)
  Both Eyes Combined: Change at Week 52 | 23.81 (17.076) | 19.87 (18.112) | 26.52 (18.341) | 23.84 (19.218) | 25.38 (19.781) | 20.37 (14.102) | 25.71 (23.057)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 41.63 (25.286) | 31.50 (18.865) | 53.57 (30.657) |  | 31.12 (24.754) | 32.22 (18.972) | 35.83 (17.546)

14. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Central Macular 2 mm Subfield EZ Partial Attenuation in the Study Eye, the Fellow Eye, and Both Eyes Combined as Measured by SD-OCT
Description: The percentage of partial attenuation of the EZ in the central macular 2 mm subfield is reported.
Time Frame: Baseline, Week 52 and Week 104
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of EZ partial attenuation
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of EZ partial attenuation
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 8.24 (10.598) | 6.09 (7.169) | 7.54 (8.630) | 6.37 (8.079) | 6.67 (7.237) | 6.93 (9.374) | 5.46 (7.746)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 18.70 (12.603) | 12.71 (13.460) | 10.96 (11.518) |  | 12.12 (11.782) | 17.09 (13.793) | 5.12 (5.509)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 6.24 (9.738) | 5.12 (9.238) | 6.73 (11.225) | 9.07 (12.589) | 9.62 (10.501) | 8.30 (12.676) | 9.17 (14.826)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 13.98 (14.829) | 7.71 (7.689) | 12.49 (18.409) |  | 12.14 (25.712) | 9.47 (17.096) | 9.30 (13.802)
  Both Eyes Combined: Change at Week 52 | 13.27 (14.756) | 9.71 (10.869) | 13.61 (15.682) | 13.96 (16.418) | 14.82 (15.686) | 13.42 (16.367) | 13.59 (17.862)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 27.52 (23.015) | 17.70 (15.710) | 22.87 (24.193) |  | 22.24 (31.056) | 24.67 (24.320) | 14.41 (14.806)

15. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Sub-RPE Central 1 mm Subfield Mean Thickness in the Study Eye, Fellow Eye and Both Eyes Combined as Measured by SD-OCT
Description: Sub-RPE compartment measures reflect the disease burden between the RPE and Bruch's membrane. The sub-RPE central 1 mm mean thickness refers to the average thickness of the retina within a 1-mm diameter circular area centered around the fovea (the central part of the retina).
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment) with both baseline and post-baseline (Week 52 and Week 104) visit sub-RPE central 1 mm subfield mean thickness data. As prespecified, data were collected and reported for participants. Hence, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
µm
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | -2.61 (5.838) | -2.89 (4.863) | -2.87 (5.842) | -0.04 (12.832) | -2.97 (5.403) | -2.13 (6.814) | 5.19 (20.081)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | -3.24 (11.423) | -4.33 (7.450) | -5.26 (9.398) |  | -3.72 (7.208) | -6.38 (9.288) | -4.72 (9.648)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | -0.84 (6.699) | -1.50 (3.274) | -2.42 (6.345) | -2.33 (8.500) | -1.13 (11.960) | -0.59 (3.463) | -5.00 (6.941)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | -3.58 (9.171) | -4.18 (6.176) | -6.73 (9.984) |  | -10.56 (11.610) | -3.90 (5.368) | -9.36 (12.776)
  Both Eyes Combined: Change at Week 52 | -3.23 (9.340) | -3.95 (5.893) | -5.05 (9.529) | -2.04 (14.876) | -3.83 (12.208) | -2.60 (7.605) | 0.40 (21.689)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | -5.74 (14.485) | -7.04 (9.644) | -11.72 (16.323) |  | -12.52 (16.342) | -9.50 (12.294) | -14.08 (21.741)

16. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Sub-RPE Central Macular 2 mm Subfield Mean Thickness in the Study Eye, Fellow Eye and Both Eyes Combined as Measured by SD-OCT
Description: Sub-RPE compartment measures reflect the disease burden between the RPE and Bruch's membrane. The sub-RPE central macular 2 mm subfield thickness refers to the thickness of the retina within a 2-mm radius in the central part of the macula.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (randomized participants who received at least 1 dose [full/partial] of study drug grouped by randomized treatment) with both baseline and post-baseline (Week 52 and Week 104) visit sub-RPE central macular 2 mm subfield mean thickness data. As prespecified, data were collected and reported for participants. Hence, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
µm
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | -2.75 (4.229) | -3.34 (3.314) | -3.02 (4.064) | -1.88 (5.550) | -3.36 (4.148) | -2.06 (3.834) | -0.15 (7.701)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | -5.80 (9.514) | -5.35 (4.290) | -6.22 (3.954) |  | -3.78 (7.190) | -4.32 (2.743) | -5.16 (4.527)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | -1.66 (4.750) | -3.07 (3.575) | -2.93 (3.552) | -3.12 (5.733) | -2.79 (7.131) | -1.24 (3.434) | -5.06 (5.370)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | -4.42 (9.773) | -9.15 (13.049) | -6.33 (5.931) |  | -9.90 (10.970) | -5.08 (2.898) | -12.30 (10.238)
  Both Eyes Combined: Change at Week 52 | -4.06 (6.749) | -5.51 (5.298) | -5.67 (5.790) | -4.50 (7.649) | -5.66 (7.552) | -3.03 (4.963) | -4.77 (9.770)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | -8.61 (12.280) | -11.28 (12.963) | -12.22 (8.602) |  | -12.03 (16.671) | -8.38 (5.509) | -17.46 (11.297)

17. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Panmacular Sub-RPE Volume in the Study Eye, Fellow Eye and Both Eyes Combined as Measured by SD-OCT
Description: Sub-RPE compartment measures reflect the disease burden between the RPE and Bruch's membrane. The panmacular sub-RPE volume refers to the total volume of fluid or space located underneath the RPE across the entire macula (the central part of the retina).
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit panmacular sub-RPE volume data. As prespecified, data were collected and reported for the participants. Therefore, the 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
mm^3
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 64 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | -0.04 (0.052) | -0.04 (0.050) | -0.05 (0.059) | -0.04 (0.066) | -0.06 (0.079) | -0.03 (0.064) | -0.03 (0.051)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 16 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | -0.08 (0.076) | -0.07 (0.085) | -0.09 (0.065) |  | -0.05 (0.094) | -0.10 (0.063) | -0.06 (0.091)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | -0.04 (0.074) | -0.04 (0.048) | -0.04 (0.054) | -0.04 (0.068) | -0.05 (0.082) | -0.02 (0.053) | -0.06 (0.062)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | -0.08 (0.084) | -0.09 (0.098) | -0.08 (0.085) |  | -0.11 (0.114) | -0.05 (0.050) | -0.17 (0.123)
  Both Eyes Combined: Change at Week 52 | -0.07 (0.102) | -0.06 (0.073) | -0.08 (0.088) | -0.08 (0.111) | -0.09 (0.142) | -0.05 (0.089) | -0.08 (0.093)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | -0.14 (0.127) | -0.12 (0.160) | -0.17 (0.128) |  | -0.14 (0.196) | -0.14 (0.085) | -0.24 (0.074)

18. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Macular Total RPE Attenuation in the Study Eye, Fellow Eye and Both Eyes Combined as Measured by SD-OCT
Description: Macular total RPE attenuation refers to the degree of thinning or loss of the RPE in the macula, the central part of the retina responsible for sharp, detailed vision. This was measured as a percentage of the macular area affected.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit macular total RPE attenuation data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: percentage of macular area
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of macular area
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 64 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 6.11 (3.874) | 5.11 (2.706) | 6.38 (3.718) | 5.48 (3.413) | 5.47 (3.043) | 5.00 (3.328) | 6.00 (3.916)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 16 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 10.66 (6.579) | 9.18 (5.951) | 11.64 (4.956) |  | 7.86 (4.673) | 12.68 (6.330) | 11.77 (5.205)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 5.23 (3.594) | 5.00 (3.549) | 5.59 (4.513) | 6.18 (4.043) | 5.55 (3.474) | 5.18 (3.740) | 7.66 (4.545)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 10.96 (6.159) | 8.50 (6.472) | 11.49 (8.582) |  | 10.38 (7.719) | 11.82 (6.691) | 16.12 (4.807)
  Both Eyes Combined: Change at Week 52 | 10.36 (6.652) | 8.58 (5.429) | 11.42 (6.976) | 10.62 (7.048) | 10.09 (6.376) | 9.06 (6.227) | 12.73 (8.186)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 18.20 (12.155) | 14.14 (11.759) | 22.52 (12.076) |  | 16.51 (12.246) | 22.14 (10.270) | 27.89 (8.760)

19. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Central 1 mm Subfield Total RPE Attenuation in the Study Eye, Fellow Eye and Both Eyes Combined as Measured by SD-OCT
Description: The percentage of total attenuation of the RPE in the central 1 mm subfield is reported.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment) with both baseline and post-baseline (Week 52 and Week 104) visit central 1 mm subfield total RPE attenuation data. As prespecified, data were collected and reported for participants. Hence, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: percentage of total RPE attenuation
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of total RPE attenuation
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 10.27 (13.204) | 8.60 (11.277) | 9.60 (13.794) | 8.16 (12.335) | 9.85 (13.381) | 9.02 (13.346) | 5.48 (9.989)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 15.56 (18.923) | 14.77 (12.017) | 19.42 (18.209) |  | 13.89 (12.330) | 28.62 (27.097) | 15.79 (29.801)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 7.48 (12.846) | 5.91 (10.333) | 8.67 (11.815) | 9.69 (15.031) | 7.33 (10.670) | 6.46 (7.800) | 14.81 (21.405)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 15.43 (13.245) | 9.84 (13.900) | 20.71 (18.542) |  | 21.88 (20.194) | 22.45 (22.899) | 23.19 (37.563)
  Both Eyes Combined: Change at Week 52 | 16.29 (21.116) | 12.79 (16.127) | 17.43 (19.549) | 16.23 (21.394) | 15.85 (19.996) | 14.08 (18.363) | 18.76 (25.857)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 26.10 (21.267) | 21.13 (18.674) | 39.11 (27.628) |  | 32.12 (28.775) | 46.58 (43.859) | 38.98 (66.640)

20. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Percent Central Macular 2 mm Subfield Total RPE Attenuation in the Study Eye, Fellow Eye and Both Eyes Combined as Measured by SD-OCT
Description: The percentage of total attenuation of the RPE in the central macular 2 mm subfield is reported.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in FAS (all randomized participants who received at least 1 dose [full/partial] of study drug grouped by randomized treatment) with both baseline and postbaseline (Week 52 and Week 104) visit central macular 2 mm subfield total RPE attenuation data. As prespecified, data were collected and reported for participants. Hence, 'Ns' reported below= number of participants analyzed regardless of which eye was evaluated. Number analyzed= participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: percentage of total RPE attenuation
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 72 | 65 | 72 | 70 | 24 | 23 | 23
percentage of total RPE attenuation
  Study Eye: Change at Week 52: number analyzed (Participants) | 69 | 65 | 72 | 68 | 23 | 23 | 22
  Study Eye: Change at Week 52 | 11.07 (8.790) | 10.86 (7.042) | 11.21 (8.539) | 10.18 (9.265) | 12.20 (9.228) | 8.89 (8.759) | 9.41 (9.869)
  Study Eye: Change at Week 104: number analyzed (Participants) | 16 | 17 | 18 | 0 | 6 | 5 | 5
  Study Eye: Change at Week 104 | 22.11 (18.777) | 20.14 (11.243) | 22.35 (9.980) |  | 14.87 (10.962) | 20.32 (5.212) | 13.47 (11.872)
  Fellow Eye: Change at Week 52: number analyzed (Participants) | 62 | 46 | 65 | 60 | 21 | 18 | 21
  Fellow Eye: Change at Week 52 | 8.84 (9.019) | 8.99 (11.116) | 10.56 (9.026) | 11.50 (8.889) | 11.30 (7.522) | 8.36 (7.234) | 14.38 (10.698)
  Fellow Eye: Change at Week 104: number analyzed (Participants) | 16 | 11 | 19 | 0 | 5 | 4 | 5
  Fellow Eye: Change at Week 104 | 17.54 (13.638) | 12.04 (10.432) | 20.96 (12.092) |  | 22.81 (19.741) | 26.77 (6.514) | 26.85 (20.134)
  Both Eyes Combined: Change at Week 52 | 18.22 (13.985) | 17.22 (13.792) | 20.75 (13.888) | 19.74 (14.674) | 21.58 (14.796) | 15.43 (11.951) | 22.13 (16.571)
  Both Eyes Combined: Change at Week 104: number analyzed (Participants) | 19 | 17 | 19 | 0 | 6 | 5 | 5
  Both Eyes Combined: Change at Week 104 | 33.38 (19.938) | 27.94 (19.154) | 42.14 (18.854) |  | 33.88 (27.642) | 41.73 (15.668) | 40.32 (28.798)

21. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Monocular Best-corrected Visual Acuity (BCVA) Scores in the Study Eye as Assessed by the Early Treatment Diabetic Retinopathy Study (ETDRS) Chart
Description: ETDRS charts present a series of five letters of equal difficulty on each row, with standardized spacing between letters and rows; there is a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Minimum score of zero, maximum score of 100. Change from baseline: a more negative score is worse outcome, a more positive score is better outcome. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome).
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit BCVA score data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 73 | 68 | 75 | 70 | 24 | 23 | 23
letters
  Change at Week 52 | -2.2 (8.56) | -2.0 (9.39) | -3.5 (11.35) | -1.8 (5.60) | -2.4 (5.74) | -2.0 (4.39) | -0.9 (6.58)
  Change at Week 104: number analyzed (Participants) | 20 | 17 | 20 | 0 | 6 | 5 | 5
  Change at Week 104 | -1.3 (4.71) | -2.2 (12.30) | -10.2 (16.37) |  | -2.7 (6.62) | -3.2 (5.54) | -5.4 (6.39)

22. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Monocular Low Luminance Visual Acuity (LLVA) Scores in the Study Eye as Assessed by the ETDRS Chart
Description: LLVA was measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. LLVA was reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Change from baseline: a negative score indicates decline in LLVA.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit LLVA score data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 74 | 67 | 72 | 70 | 24 | 23 | 22
letters
  Change at Week 52 | -6.3 (11.61) | -4.6 (11.77) | -4.0 (11.23) | -4.8 (15.96) | -7.7 (13.43) | -1.2 (17.90) | -5.5 (16.71)
  Change at Week 104: number analyzed (Participants) | 44 | 41 | 49 | 0 | 13 | 14 | 12
  Change at Week 104 | -10.3 (14.27) | -9.9 (14.15) | -8.9 (10.39) |  | -8.0 (10.37) | -3.9 (20.88) | -11.8 (15.86)

23. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in Low Luminance Deficit (LLD) (BCVA-LLVA) Score in the Study Eye
Description: LLD score was calculated as the difference between BCVA and LLVA (BCVA-LLVA) scores. BCVA and LLVA were reported as the number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision. LLD is a measure of visual acuity impairment in low-light conditions. A higher LLD score indicates a greater difference between vision in bright and dim light, suggesting a more significant loss of visual function in low-luminance settings.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit LLD score data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 74 | 67 | 71 | 70 | 24 | 23 | 22
letters
  Change at Week 52 | 4.3 (13.30) | 2.6 (13.68) | 0.3 (15.67) | 2.9 (15.18) | 5.3 (12.56) | -0.8 (17.15) | 4.5 (15.84)
  Change at Week 104: number analyzed (Participants) | 44 | 41 | 48 | 0 | 13 | 14 | 12
  Change at Week 104 | 5.6 (17.11) | 6.3 (15.22) | 0.5 (19.93) |  | 4.4 (13.83) | -2.7 (24.00) | 9.3 (15.91)

24. Secondary Outcome: Change From Baseline to Week 52 And Week 104 in Monocular Reading Speeds in the Study Eye as Assessed by Minnesota Low Vision Reading Test (MNRead) Acuity Charts or Radner Reading Charts
Description: MNRead acuity cards were continuous-text reading-acuity cards suitable for measuring the reading acuity and reading speed of normal and low-vision participants. The MNRead acuity cards consisted of single, simple sentences with equal numbers of characters. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. The Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. The reading test was stopped when the reading time was longer than 20 seconds or when the participant was making severe errors. A negative change from baseline indicates a decrease in the monocular reading speed; disease worsening.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit reading speed data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: words per minute (wpm)
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 67 | 62 | 58 | 56 | 20 | 15 | 20
words per minute (wpm)
  Change at Week 52 | -137.36 (1016.889) | -19.80 (42.134) | -13.47 (77.927) | -14.55 (81.313) | 16.22 (104.097) | -41.54 (53.752) | -30.46 (61.042)
  Change at Week 104: number analyzed (Participants) | 39 | 37 | 35 | 0 | 9 | 10 | 9
  Change at Week 104 | 16.04 (142.422) | -23.70 (57.745) | -29.01 (65.896) |  | -59.41 (43.156) | 30.18 (144.094) | -47.13 (71.218)

25. Secondary Outcome: Change From Baseline to Week 52 and Week 104 in National Eye Institute Visual Function Questionnaire (NEI VFQ-25) Composite Scores
Description: The NEI VFQ-25 instrument measures dimensions of self-reported vision-targeted health status of individuals with chronic eye conditions. The NEI VFQ-25 consists of 11 vision related domains: global vision rating, difficulty with near vision activities, difficulty with distance vision activities, limitations in social function related to vision, role limitations, dependency on others due to vision, mental health symptoms due to vision, driving difficulties, limitations with peripheral- and color-vision, and ocular pain. The NEI VFQ-25 also includes a single item measuring general health. A composite score averages the vision related domains and ranges from 0 (worse) to 100 (best). A higher score represents better functioning. A negative change from baseline indicates a decrease in the visual functioning; disease worsening.
Time Frame: Baseline, Week 52 and Week 104
Population: All participants in the FAS (all randomized participants who received at least 1 dose [full or partial] of study drug grouped by randomized treatment group) with both baseline and post-baseline (Week 52 and Week 104) visit NEI VFQ-25 scores data. As prespecified, data were collected and reported for participants. Therefore, 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated. Number analyzed = participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo | Placebo - Danicopan 100 mg BID | Placebo - Danicopan 200 mg BID | Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 73 | 67 | 75 | 70 | 24 | 23 | 23
units on a scale
  Change at Week 52 | -0.425 (9.6019) | -5.816 (11.9162) | -4.456 (9.4963) | -1.578 (11.0757) | -1.058 (9.1822) | -4.856 (11.4575) | 1.156 (12.0823)
  Change at Week 104: number analyzed (Participants) | 31 | 29 | 34 | 0 | 9 | 8 | 9
  Change at Week 104 | -7.676 (16.3251) | -8.478 (13.5192) | -7.454 (14.2207) |  | -0.332 (13.3618) | 0.535 (10.7239) | -9.944 (13.4043)

26. Secondary Outcome: Plasma Concentration of Danicopan
Description: All values below the limit of quantification (<0.1 nanograms [ng]/milliliter [mL]) were set to 0 for calculation of summary statistics.
Time Frame: Day 1 and Week 52
Population: Pharmacokinetic (PK) Analysis Set included all participants who received at least 1 dose (full or partial) of study drug and had at least 1 measurable concentration value. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD
Number analyzed (Participants) | 91 | 87 | 89
ng/mL
  Day 1: Predose | 0.4 (3.41) | 0 (0) | 0.2 (1.67)
  Day 1: 2 Hour Postdose: number analyzed (Participants) | 90 | 85 | 88
  Day 1: 2 Hour Postdose | 289.6 (202.88) | 507.5 (279.71) | 844.5 (563.54)
  Week 52: Predose: number analyzed (Participants) | 70 | 67 | 72
  Week 52: Predose | 62.5 (40.64) | 127.7 (100.78) | 88.1 (138.95)
  Week 52: 2 Hour Postdose: number analyzed (Participants) | 72 | 65 | 72
  Week 52: 2 Hour Postdose | 381.6 (219.22) | 704.4 (336.37) | 919.5 (709.94)

27. Secondary Outcome: Change From Baseline in Ex Vivo Serum Alternative Pathway (AP) Activity
Description: Serum AP functional activity was measured by the Wieslab functional immunoassay method.
Time Frame: Week 52 (pre-dose, 2 hours post-dose)
Population: Pharmacodynamic (PD) Analysis Set included all participants who received at least 1 dose (full or partial) of study drug and had at least 1 measurable PD value. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of activity
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo
Number analyzed (Participants) | 67 | 68 | 70 | 68
percentage of activity
  Change at Week 52: Predose: number analyzed (Participants) | 64 | 68 | 68 | 68
  Change at Week 52: Predose | -5.9 (17.49) | -21.3 (29.90) | -8.2 (24.48) | 2.7 (17.12)
  Change at Week 52: 2 Hour Postdose: number analyzed (Participants) | 67 | 62 | 70 | 64
  Change at Week 52: 2 Hour Postdose | -58.5 (27.85) | -75.3 (23.17) | -74.8 (28.82) | -23.1 (42.12)

28. Secondary Outcome: Change From Baseline in Plasma Bb Fragment of Complement Factor B (Bb) Concentration
Time Frame: Baseline, Week 52 (pre-dose)
Population: PD Analysis Set included all participants who received at least 1 dose (full or partial) of study drug and had at least 1 measurable PD value. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Danicopan 100 mg BID | Danicopan 200 mg BID | Danicopan 400 mg QD | Placebo
Number analyzed (Participants) | 66 | 65 | 72 | 70
µg/mL | -0.3 (0.77) | -0.7 (0.94) | -0.2 (0.55) | -0.1 (0.55)

29. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Events Leading To Discontinuation of Study Drug Throughout the Study
Description: An adverse event (AE) was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), or an important medical event or reaction. A TEAE was defined as any AE that started during or after the first dose of study intervention. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 through Week 108
Population: Safety Set included all participants who received at least 1 dose (full or partial) of study drug grouped by treatment actually received. As prespecified, data were collected and reported for the participants. Therefore, the 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Evaluation Period: Danicopan 100 mg BID: Participants received danicopan 100 mg BID during the 52-week Primary Evaluation Period.
- Primary Evaluation Period: Danicopan 200 mg BID: Participants received danicopan 200 mg BID during the 52-week Primary Evaluation Period.
- Primary Evaluation Period: Danicopan 400 mg QD: Participants received danicopan 400 mg QD during the 52-week Primary Evaluation Period.
- Primary Evaluation Period: Placebo: Participants received matching placebo during the 52-week Primary Evaluation Period.
- Secondary Evaluation Period: Danicopan 100 mg BID: Participants received danicopan 100 mg BID during the 52-week Secondary Evaluation Period.
- Secondary Evaluation Period: Danicopan 200 mg BID: Participants received danicopan 200 mg BID during the 52-week Secondary Evaluation Period.
- Secondary Evaluation Period: Danicopan 400 mg QD: Participants received danicopan 400 mg QD during the 52-week Secondary Evaluation Period.
- Secondary Evaluation Period: Placebo - Danicopan 100 mg BID: Participants who received placebo during the primary evaluation period (up to Week 52), were re-randomized to receive danicopan 100 mg BID for the remainder of the study.
- Secondary Evaluation Period: Placebo - Danicopan 200 mg BID: Participants who received placebo during the primary evaluation period (up to Week 52), were re-randomized to receive danicopan 200 mg BID for the remainder of the study.
- Secondary Evaluation Period: Placebo - Danicopan 400 mg QD: Participants who received placebo during the primary evaluation period (up to Week 52), were re-randomized to receive danicopan 400 mg QD for the remainder of the study.
Arm/Group | Primary Evaluation Period: Danicopan 100 mg BID | Primary Evaluation Period: Danicopan 200 mg BID | Primary Evaluation Period: Danicopan 400 mg QD | Primary Evaluation Period: Placebo | Secondary Evaluation Period: Danicopan 100 mg BID | Secondary Evaluation Period: Danicopan 200 mg BID | Secondary Evaluation Period: Danicopan 400 mg QD | Secondary Evaluation Period: Placebo - Danicopan 100 mg BID | Secondary Evaluation Period: Placebo - Danicopan 200 mg BID | Secondary Evaluation Period: Placebo - Danicopan 400 mg QD
Number analyzed (Participants) | 93 | 91 | 91 | 90 | 73 | 67 | 73 | 24 | 23 | 23
Participants
  Any TEAEs | 79 | 83 | 76 | 71 | 51 | 37 | 46 | 19 | 12 | 17
  SAEs | 14 | 19 | 16 | 15 | 8 | 10 | 8 | 6 | 4 | 4
  Events Leading To Discontinuation of Study Drug | 11 | 15 | 9 | 11 | 1 | 2 | 4 | 0 | 2 | 4

ADVERSE EVENTS:
Time Frame: Day 1 through Week 108
Description: Safety Set included all participants who received at least 1 dose (full or partial) of study drug grouped by treatment actually received. 'Deaths' as the 'reason for study discontinuation' have been reported in the participant flow section and 'all deaths' have been reported in the 'All-cause mortality' section.
  As prespecified, data were collected and reported for the participants. Therefore, the 'Ns' reported below = number of participants analyzed regardless of which eye was evaluated.
Arm/Group | Primary Evaluation Period: Danicopan 100 mg BID | Primary Evaluation Period: Danicopan 200 mg BID | Primary Evaluation Period: Danicopan 400 mg QD | Primary Evaluation Period: Placebo | Secondary Evaluation Period: Danicopan 100 mg BID | Secondary Evaluation Period: Danicopan 200 mg BID | Secondary Evaluation Period: Danicopan 400 mg QD | Secondary Evaluation Period: Placebo - Danicopan 100 mg BID | Secondary Evaluation Period: Placebo - Danicopan 200 mg BID | Secondary Evaluation Period: Placebo - Danicopan 400 mg QD
All-Cause Mortality (participants affected / at risk) | 0/93 | 1/91 | 0/91 | 3/90 | 1/73 | 1/67 | 1/73 | 1/24 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 14/93 | 19/91 | 16/91 | 15/90 | 8/73 | 10/67 | 8/73 | 6/24 | 4/23 | 4/23
Other Adverse Events (participants affected / at risk) | 44/93 | 42/91 | 33/91 | 33/90 | 22/73 | 14/67 | 16/73 | 12/24 | 7/23 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Evaluation Period: Danicopan 100 mg BID (N=93) | Primary Evaluation Period: Danicopan 200 mg BID (N=91) | Primary Evaluation Period: Danicopan 400 mg QD (N=91) | Primary Evaluation Period: Placebo (N=90) | Secondary Evaluation Period: Danicopan 100 mg BID (N=73) | Secondary Evaluation Period: Danicopan 200 mg BID (N=67) | Secondary Evaluation Period: Danicopan 400 mg QD (N=73) | Secondary Evaluation Period: Placebo - Danicopan 100 mg BID (N=24) | Secondary Evaluation Period: Placebo - Danicopan 200 mg BID (N=23) | Secondary Evaluation Period: Placebo - Danicopan 400 mg QD (N=23)
Macular hole (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Induration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Superinfection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neovascular age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic foot infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Evaluation Period: Danicopan 100 mg BID (N=93) | Primary Evaluation Period: Danicopan 200 mg BID (N=91) | Primary Evaluation Period: Danicopan 400 mg QD (N=91) | Primary Evaluation Period: Placebo (N=90) | Secondary Evaluation Period: Danicopan 100 mg BID (N=73) | Secondary Evaluation Period: Danicopan 200 mg BID (N=67) | Secondary Evaluation Period: Danicopan 400 mg QD (N=73) | Secondary Evaluation Period: Placebo - Danicopan 100 mg BID (N=24) | Secondary Evaluation Period: Placebo - Danicopan 200 mg BID (N=23) | Secondary Evaluation Period: Placebo - Danicopan 400 mg QD (N=23)
Neovascular age-related macular degeneration (Eye disorders) | 5 | 5 | 5 | 3 | 3 | 2 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 4 | 3 | 3 | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 5 | 7 | 9 | 8 | 2 | 3 | 6 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 6 | 6 | 9 | 5 | 8 | 2 | 4 | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 9 | 5 | 3 | 8 | 4 | 3 | 3 | 2 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 9 | 7 | 5 | 3 | 1 | 1 | 0 | 3 | 2 | 3
C-reactive protein increased (Investigations) | 1 | 3 | 7 | 6 | 3 | 2 | 2 | 3 | 0 | 1
Hepatic enzyme increased (Investigations) | 5 | 6 | 4 | 0 | 1 | 0 | 0 | 1 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 4 | 4 | 5 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 5 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 5 | 4 | 6 | 2 | 1 | 1 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 6 | 4 | 3 | 3 | 1 | 4 | 2 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 3 | 1 | 3 | 0 | 3 | 4 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 3 | 6 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 2 | 1 | 2 | 1 | 0 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early because the primary efficacy endpoint was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT05019521/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT05019521/SAP_001.pdf